CLINICAL TRIAL: NCT01169545
Title: Cancer, Vulnerability, and Financial Quality of Life: A Mixed Methods Study
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Christine Callahan, PhD, LCSW-C, clinical social worker and PhD candidate, Georgetown University
Other Study IDs: 2010-090
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Cancer
Keywords: any type of cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer patients over the age of 18: Cancer patients over the age of 18 who are receiving active treatment.

SUMMARY:
The primary purpose of this study is to examine how vulnerabilities in psychological and social situations affect financial quality of life.

DETAILED DESCRIPTION:
The primary purpose of this study is to examine how vulnerabilities in psychological and social situations affect financial quality of life. For people who are experiencing financial hardship, a cancer diagnosis can be devastating. For others, cancer may cause or even worsen financial stress, for example, with their work, their ability to maintain benefits such as health insurance, their ability to pay bills, and their ability to get the cancer treatment they need. The impact of cancer on financial quality of life is an important area of study within cancer care. Considering the financial burden of cancer also lends greater appreciation for the problems that people face if they cannot handle cancer's costs, or if needed resources are either not present or are too stretched to help with the care they need. For this study, up to 180 cancer patients will be interviewed with a written questionnaire. Of this group, 15 people will also be asked if they would like to participate in a follow-up personal interview with the researcher. The major hypothesis of this study is: The greater the vulnerabilities in predisposing factors and enabling factors, the greater the need factors with respect to cancer diagnosis and treatment, and the lower the perceived ability to adhere to treatment, the poorer will be the financial quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Any cancer patient over the age of 18 who can speak and understand English and can provide informed consent

Exclusion Criteria:

* Pediatric patients; non-English-speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any cancer patient over the age of 18 who can speak and understand English and can provide informed consent
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Identification of Potential Vulnerabilities | May 2010 to October 2012
  To examine how vulnerabilities in psychological and social situations affect financial quality of life. The dependent variable in this study is financial quality of life, defined as the ability to manage all current and future (including unexpected) financial obligations related to cancer care, within the context of sound health-care decision-making. Under the theoretical framework used, the first three independent variables selected under the predisposing domain are housing instability, personal control within the larger context of health locus of control, and demographics. Under the enabling domain, the next variables measured are income and financial stress, presence of health insurance and health insurance adequacy, perceived barriers to care, and social support. For the need domain, a patient's experience with cancer in terms of treatment and acuity are measured. Variables are measured using standardized instruments or in the absence of one, a scale composed by the researcher.

CONTACTS AND LOCATIONS:
Overall Officials: Christine C. Callahan, MSW, Principal Investigator — The Catholic University of America